CLINICAL TRIAL: NCT04111302
Title: Cohort Study of Auricular Pressure Therapy for Intervention of Postoperative Pain of Hemorrhoidectiomy
Brief Title: Cohort Study of Auricular Acupressure for Postoperative Pain After Hemorrhoidectiomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CXTD1702
Record Dates: First submitted 2019-09-17; First posted 2019-10-01 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain After Hemorrhoidectomy
Keywords: hemorrhoidectiomy; postoperative pain; auricular pressure
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IV-PCA (Experimental): use IV-PCA for postoperative pain
  Interventions: Other: IV-PCA
- IV-dezocine (Experimental): use IV-dezocine for postoperative pain
  Interventions: Other: IV-dezocine
- IV-PCA+AA (Experimental): use IV-PCA and AA for postoperative pain
  Interventions: Other: IV-PCA+AA
- IV-dezocine+AA (Experimental): use IV-dezocine and AA for postoperative pain
  Interventions: Other: IV-dezocine+AA

INTERVENTIONS:
Other: IV-PCA — IV-PCA contains dezocine 10mg, sufentanil 100ug, metoclopramide 20mg and normal saline are prepared into 100ml solution and pumped evenly at the speed of 2ml/h.
  Arms: IV-PCA
Other: IV-dezocine — IV-dezocine contains dezocine 5mg and 250ml normal saline are made into solution and injected intravenously twice a day for 3 consecutive days after surgery.
  Arms: IV-dezocine
Other: IV-PCA+AA — IV-PCA contains dezocine 10mg, sufentanil 100ug, metoclopramide 20mg and normal saline are prepared into 100ml solution and pumped evenly at the speed of 2ml/h. And selecting the auricular points TF4, AH6a, HX2, HX5, CO4, AT4 and cowherb seeds will be attached to each auricular point after the auricle skin is disinfected. The participants will be asked to press the cowherb seeds against the auricular points every 2 hours during waking hours; each point is stimulated for one minute. Auricular points are pressed unilaterally, and the cowherb seeds will be replaced with new ones every 2 days, alternating from left to right.
  Arms: IV-PCA+AA
Other: IV-dezocine+AA — IV-dezocine contains dezocine 5mg and 250ml normal saline are made into solution and injected intravenously twice a day for 3 consecutive days after surgery.And selecting the auricular points TF4, AH6a, HX2, HX5, CO4, AT4 and cowherb seeds will be attached to each auricular point after the auricle skin is disinfected. The participants will be asked to press the cowherb seeds against the auricular points every 2 hours during waking hours; each point is stimulated for one minute. Auricular points are pressed unilaterally, and the cowherb seeds will be replaced with new ones every 2 days, alternating from left to right.
  Arms: IV-dezocine+AA

SUMMARY:
Auricular pressure is effective for postoperative analgesia after hemorrhoidectomy, but the evidence is not sufficient.

DETAILED DESCRIPTION:
This is a cohort study to study the analgesic effect of auricular pressure pill on persistent pain after hemorrhoidectiomy. Baseline pain intensity scores (VAS>3) of the subjects will be collected 3 hours after the operation of the patients. By doctors' recommend interventions and the patients' preference, eligible subjects were naturally divided into the following queues: intravenous patient-controlled analgesia(IV-PCA),intravenous dezocine(IV-dezocine),intravenous patient-controlled analgesia+auricular acupressure(IV-PCA+AA),intravenous dezocine+auricular acupressure(IV-dezocine+AA). The treatment will last 5-7 days. Participants will receive auricular pressure once two days, and receive VAS, concomitant medication, PONV intensity scale and peripheral edema were recorded daily, and after the operation 3 hours, 3 days and 7 days the patients will receive anxiety and depression scale(HAD) , and VAS data will be collected by telephone at 3 and 6 months after the operation.

The main indicators will be analyzed by VAS score and generalized linear model, with VAS results as the dependent variable, grouping as the random factor, surgical method, mixed hemorrhoid classification as fixed effects factor, and age, course of disease, baseline VAS scores and VAS follow-up time point as the covariables to analysis VAS score improved relations between various factors. Analgesic usage, ease pain evaluation method and using the same scale and HAD GLM model analysis.The secondary indicator analgesic usage rate will be analyzed using logistic regression analysis. fixed effects and covariate factors set with the GLM model.

The purpose of this study was to seek high quality evidence-based medical evidence for intervention of auricular pressure pills on postoperative pain of hemorrhoidectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of grade II-IV mixed hemorrhoids and meet the operation conditions;
2. Age 18~65;
3. External stripping and internal ligation of mixed hemorrhoids, general anesthesia or lumbar shu point anesthesia;
4. VAS score ≥3 points;
5. Sign informed consent.

Exclusion Criteria:

* Combined cognitive impairment could not complete the efficacy evaluation;
* With other gastrointestinal conditions found during operation;
* With severe cardiovascular, hepatic, or renal diseases;
* With opioid addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale(VAS) | Day 1 to 7 and month 3 and 6 after natural allocation
  It is a unidimensional measure providing a simple solution for measuring subjective experience. The VAS scale is a 10-cm line with 0 cm indicating no symptoms and 10 cm indicates the greatest extent of symptoms.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression scale(HAD) | Three hours, day 3, and day 7 after natural allocation
  The HAD scale included measures of anxiety and depression, with scores ranging from 0 to 21. 0-7 points means asymptomatic;A score of 8-10 means suspicious;A score of 11 to 21 means definitely symptomatic( anxiety or depression).

OTHER OUTCOMES:
The utilization rate of analgesic drugs（Diclofenac Sodium Dual Release Enteric-coated Capsules) | Day 7 after natural allocation
  The ratio of patients using analgesic drugs in each group was calculated (Patients who take bisphenolics once are considered users), and the utilization rate = number of users/total number of users ×100%.
Amount of analgesic drugs (Diclofenac Sodium Dual Release Enteric-coated Capsules) | Day 7 after natural allocation
  The total analgesic drugs dose of each group was considered as the amount of analgesics in the group
Tissue edema | Day 3,day 4,day 5,day 6 and day 7 after natural allocation
  The degree of tissue edema was observed and recorded truthfully

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zheng, phD, Principal Investigator — Chengdu University of Traditional Chinese Medicine